CLINICAL TRIAL: NCT01175603
Title: Preventing Postpartum Depression in African American Home Visiting Clients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Abell Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHMI ICTR 2009; ICTR 2009 (Other: Johns Hopkins University ICTR)
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Depression
Keywords: depression, African American, home visiting, prevention
MeSH Terms: conditions — Depression | interventions — Acclimatization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral intervention (Experimental): Women in the intervention condition will receive 6 two-hour intervention sessions delivered weekly in a group format by the Study Clinician. Each session contains didactic instruction on core content, as well as activities and group discussion. One of the strengths of embedding the MB Course within home visiting is our ability to have home visitors reinforce the material presented by the Study Clinician. The 6-week curriculum is divided into three modules: (a) pleasant activities, (b) thoughts, and (c) relationships with others. Each module has two sessions. These sessions map onto core cognitive-behavioral concepts.
  Interventions: Behavioral: Mothers and Babies Course (Adapted for Baltimore Home Visiting Programs)
- Usual home visiting (No Intervention): Women in the control group will receive usual home visiting services and information on postpartum depression.

INTERVENTIONS:
Behavioral: Mothers and Babies Course (Adapted for Baltimore Home Visiting Programs) — 6 weekly 2-hour cognitive-behavioral intervention sessions held in group format
  Arms: Cognitive behavioral intervention

SUMMARY:
The goal of this study is to determine whether a 6 week intervention is effective in preventing the worsening of depressive symptoms and development of clinical depression in low-income African American pregnant and recently delivered women who are enrolled in home visiting programs.

DETAILED DESCRIPTION:
This study will conduct a randomized controlled trial (RCT) with women from four Baltimore City home visiting programs. We will screen 200 women who are pregnant or have a child < 6 months for study inclusion; 91 women at elevated risk for developing postpartum depression (PPD) will be randomized to an intervention (MB Course) or usual home visiting control group. Women in the intervention group will receive the 6-week MB Course delivered in a group setting by the Study Clinician with reinforcing messages provided by home visitors during 1-on-1 home visits, while women in the attention control will receive usual home visiting services and information on postpartum depression. Primary outcomes include depressive symptoms and depressive episodes.

ELIGIBILITY:
Inclusion Criteria:

* pregnant or has child < 6 months of age
* enrolled in home visiting program
* exhibiting elevated depressive symptoms and/or personal history of clinical depression

Exclusion Criteria:

* no current clinical depression at time of enrollment

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Baseline
Depressive symptoms | 1 week post intervention
Depressive Symptoms | 3 months post-intervention
Depressive symptoms | 6 months post-intervention

SECONDARY OUTCOMES:
Depressive episodes | 3 months post-intervention
Depressive Episodes | 6 Months Post-Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shiv D Tandon, PhD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - People's Community Health Center, Baltimore, Maryland
  - DRUM Healthy Families, Baltimore, Maryland
  - Maternal and Infant Nursing Program, Baltimore, Maryland
  - Sinai Hospital Perinatal Depression Outreach Program, Baltimore, Maryland